CLINICAL TRIAL: NCT00447694
Title: An Open Label Trial Evaluating Cardiac T2* in Beta-thalassemia Patients on Deferasirox (ICL670) Treatment for 18 Months
Brief Title: Cardiac T2* in Beta-thalassemia Patients on Deferasirox Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670AUS04
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Beta-thalassemia; Iron Overload
Keywords: Iron Chelation; Deferasirox; Chelator; Desferal; beta-thalassemia; Iron overload
MeSH Terms: conditions — beta-Thalassemia; Iron Overload | interventions — Deferasirox

ARMS (1):
- deferasirox every day for 77 weeks (Experimental): Participants received Deferasirox 30 milligrams per kilogram per day (mg/kg/day) orally once daily (OD), 30 minutes before breakfast, preferably around the same time every morning if possible. Deferasirox tablets were dropped into water or orange juice, or apple juice and stirred until completely dispersed. For doses less than 1 gram (g), tablets were dissolved in at least 100 milliliter (mL) of liquid; for doses of 1 to 3 g, tablets were dissolved in at least 200 mL. After tablets were fully disintegrated, the liquid was promptly consumed.
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox — Oral deferasirox 30mg/kg/day once per day for 77 weeks.

SUMMARY:
The purpose of this trial is to evaluate changes in cardiac iron as measured by MRI T2* in beta-thalassemia patients with deferasirox treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female β-thalassemia outpatients on chronic transfusion therapy (defined as > 8 transfusions per year)
* Lifetime minimum of 100 previous packed red blood cell transfusions
* Patients currently on chelation therapy will require a one day wash out prior to the first dose of study drug
* Age ≥ 10 years
* Sexually active females of childbearing potential must have a negative serum or urine pregnancy test and use an effective method of contraception, or must have undergone clinically documented total hysterectomy.

Exclusion Criteria:

* Ejection Fraction < 56 % measured using steady-state free precession imaging by MRI
* Contraindication to MRI, including cardiac pacemaker, brain aneurysm clip, implanted neurostimulator, insulin pump, cochlear implant, metal slivers in the eyes, intrauterine device or any other MRI incompatible metal implants or intractable claustrophobia
* Abnormal laboratory values as defined by the protocol
* Clinical or laboratory evidence of active Hepatitis B or Hepatitis C
* History of HIV positive test result (ELISA or Western blot)
* Uncontrolled systemic hypertension
* Second or third degree A-V block
* Life-threatening arrhythmias, including sustained ventricular tachycardia and aborted sudden death, within the last year
* History of cardiac conditions or unstable cardiac disease not controlled by standard medical therapy
* History of clinically relevant ocular toxicity related to iron chelation
* Systemic diseases (cardiovascular, renal, hepatic, etc.) which would prevent study treatment
* Pregnancy or breast feeding (documented negative pregnancy test required for study entry)
* Patients enrolled in an ongoing clinical trial of deferasirox (ICL670) cannot be withdrawn in order to participate in this study
* Treatment with systemic investigational drug within the past 4 weeks or topical investigational drug within the past 7 days
* Other surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of any drug
* History of non-compliance to medical regimens or patients who are considered potentially unreliable and/or not cooperative
* Other inclusion/exclusion criteria may apply

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Coates, MD, Principal Investigator — Childresn's Hospital of Los Angeles; Alexis Thompson, MD, Principal Investigator — Children's Memorial Hospital of Chicago; Paul Harmatz, MD, Principal Investigator — Children's Hospital and Research Center at Oakland
Locations (3):
- United States (3):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Children's Memorial Hospital, Chicago, Illinois

REFERENCES:
- [Derived] Wood JC, Glynos T, Thompson A, Giardina P, Harmatz P, Kang BP, Paley C, Coates TD. Relationship between labile plasma iron, liver iron concentration and cardiac response in a deferasirox monotherapy trial. Haematologica. 2011 Jul;96(7):1055-8. doi: 10.3324/haematol.2010.032862. Epub 2011 Mar 10. PMID 21393329
- [Derived] Wood JC, Kang BP, Thompson A, Giardina P, Harmatz P, Glynos T, Paley C, Coates TD. The effect of deferasirox on cardiac iron in thalassemia major: impact of total body iron stores. Blood. 2010 Jul 29;116(4):537-43. doi: 10.1182/blood-2009-11-250308. Epub 2010 Apr 26. PMID 20421452
- See also: Novartis Clinical Trial results website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=3642

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 4 centers in the United States
Pre-assignment Details: A total number of participants planned for this study was 30. The total number of 28 participants enrolled in the study, of these 22 completed the study and 6 discontinued the study.
Groups:
- Deferasirox: Participants received Deferasirox 30 milligrams per kilogram per day (mg/kg/day) orally once daily (OD), 30 minutes before breakfast, preferably around the same time every morning if possible. Deferasirox tablets were dropped into water or orange juice, or apple juice and stirred until completely dispersed. For doses less than 1 gram (g), tablets were dissolved in at least 100 milliliter (mL) of liquid; for doses of 1 to 3 g, tablets were dissolved in at least 200 mL. After tablets were fully disintegrated, the liquid was promptly consumed.
Period: Overall Study
Arm/Group | Deferasirox
Started | 28
Completed | 22
Not Completed | 6
Not completed — Adverse Event | 2
Not completed — Abnormal laboratory value | 1
Not completed — Abnormal test procedure result | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: The analysis was performed in Intent-to-treat (ITT) population, defined as all enrolled participants who received at least 1 dose of study drug and had at least 1 post-baseline assessment.
Groups:
- Deferasirox: Participants received Deferasirox 30 mg/kg/day orally OD, 30 minutes before breakfast, preferably around the same time every morning if possible. Deferasirox tablets were dropped into water or orange juice, or apple juice and stirred until completely dispersed. For doses less than 1 g, tablets were dissolved in at least 100 mL of liquid; for doses of 1 to 3 g, tablets were dissolved in at least 200 mL. After tablets were fully disintegrated, the liquid was promptly consumed.
Arm/Group | Deferasirox
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.6 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 8
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 9
  Black | 0
  Oriental | 7
  Other | 12

OUTCOME MEASURES:

1. Primary Outcome: Magnetic Resonance Imaging (MRI) T2* and Absolute Change From Baseline in MRI T2*
Description: Cardiac T2* was measured in the short axis plane at the widest point of a 4-chamber localizer using custom breath-hold R2* gradient echo sequences modeled after techniques used by Anderson et al (2001) and Westwood et al (2003).
Time Frame: From Baseline to 25, 49, 77 Week
Population: The analysis was performed in Completer population (CP) consists of those participants who had a Week 77 MRI.
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | Deferasirox
Number analyzed (Participants) | 22
milliseconds (msec)
  Baseline | 9.92 (3.922)
  Week 25: number analyzed (Participants) | 21
  Week 25 | 11.73 (6.091)
  Week 25 Absolute Change from Baseline: number analyzed (Participants) | 21
  Week 25 Absolute Change from Baseline | 1.77 (3.203)
  Week 49 | 11.93 (6.489)
  Week 49 Absolute Change from Baseline | 2.01 (3.792)
  Week 77 | 12.10 (6.461)
  Week 77 Absolute Change from Baseline | 2.18 (3.927)

2. Secondary Outcome: Change From Baseline in Liver Iron Concentration (LIC) Was Measured by MRI R2 From Absolute Change From Baseline to 101 Weeks
Description: MRI evaluation of liver iron concentration has been validated by liver biopsy (St Pierre et al 2005). Studies comparing T2* values of liver iron concentration (LIC) with LIC as assessed by biopsy have confirmed that T2* values reflect liver iron content (Wood et al 2003b). Direct tissue-validation of cardiac T2* measurements in humans has not been performed because endomyocardial biopsy is a dangerous and unreliable indicator of cardiac iron overload (Olson et al 1989, Fitchett et al 1980). However, it has been shown that cardiac T2* accurately reflects cardiac iron in a gerbil iron cardiomyopathy model (Wood et al 2004b). T2* measurements have shown excellent inter-scanner and inter-exam reproducibility, making them suitable for longitudinal monitoring (Westwood et al 2003a, Westwood et al 2003b).
Time Frame: From Baseline to 25, 49, 77 Week
Population: The analysis was performed in Completer population consists of those participants who had a Week 77 MRI.
Measure: Mean (Standard Deviation); unit: mg Fe/g dw liver
Arm/Group | Deferasirox
Number analyzed (Participants) | 22
mg Fe/g dw liver
  Baseline | 19.85 (3.309)
  Week 25: number analyzed (Participants) | 21
  Week 25 | 17.23 (15.393)
  Week 25 Absolute Change from Baseline: number analyzed (Participants) | 21
  Week 25 Absolute Change from Baseline | -2.89 (4.169)
  Week 49 | 17.0 (17.548)
  Week 49 Absolute Change from Baseline | -2.85 (4.883)
  Week 77 | 16.62 (20.114)
  Week 77 Absolute Change from Baseline | -3.23 (7.708)

3. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF) and Change in Left Ventricular Ejection Fraction From Baseline to 101 Weeks
Description: Magnetic resonance imaging (MRI)-measured cardiac T2* and cardiac function reflected by left and right ventricle ejection fraction. A standardized MRI protocol for T2* acquisition technique will be used in the centers. Images will be reviewed centrally by an expert MRI reader.
Time Frame: From Baseline to 25, 49, 77 Week
Population: The analysis was performed in Completer population consisting of those participants who had a Week 77 MRI.
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 22
percentage of participants
  Baseline: number analyzed (Participants) | 21
  Baseline | 64.01 (6.751)
  Week 25: number analyzed (Participants) | 21
  Week 25 | 62.17 (6.352)
  Week 25 Absolute change from baseline: number analyzed (Participants) | 21
  Week 25 Absolute change from baseline | -1.84 (7.306)
  Week 49 | 61.61 (13.726)
  Week 49 Absolute change from baseline: number analyzed (Participants) | 21
  Week 49 Absolute change from baseline | -2.68 (14.546)
  Week 77 | 63.84 (6.112)
  Week 77 Absolute change from baseline: number analyzed (Participants) | 21
  Week 77 Absolute change from baseline | 0.11 (7.299)

4. Secondary Outcome: Serum Ferritin and Changes From Baseline in Serum Ferritin During Study
Description: Serum ferritin will be assessed at each study visit. Analysis was performed in Completer population consists of those participants who had a Week 77 MRI.
Time Frame: From Baseline to 25, 49, 77 Week
Population: The analysis was performed in Completer population consists of those participants who had a Week 77 MRI.
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Deferasirox
Number analyzed (Participants) | 22
μg/L
  Baseline | 4343.75 (3486.525)
  Week 25 | 4280.77 (5261.563)
  Week 25 Absolute change from baseline | -62.98 (2294.635)
  Week 49: number analyzed (Participants) | 21
  Week 49 | 3759.29 (3966.107)
  Week 49 Absolute change from baseline: number analyzed (Participants) | 21
  Week 49 Absolute change from baseline | -593.36 (1534.040)
  Week 77: number analyzed (Participants) | 21
  Week 77 | 3179.81 (3439.357)
  Week 77 Absolute change from baseline: number analyzed (Participants) | 21
  Week 77 Absolute change from baseline | -882.74 (1368.202)

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All adverse events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit (LPLV) up to week 77.
Description: The analysis was performed on safety set population defined as all participants who received study drug and had at least one post-baseline safety assessment.
Groups:
- All Patients: Participants received Deferasirox 30 mg/kg/day orally OD, 30 minutes before breakfast, preferably around the same time every morning if possible. Deferasirox tablets were dropped into water or orange juice, or apple juice and stirred until completely dispersed. For doses less than 1 g, tablets were dissolved in at least 100 mL of liquid; for doses of 1 to 3 g, tablets were dissolved in at least 200 mL. After tablets were fully disintegrated, the liquid was promptly consumed.
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 8/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=27)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Fanconi syndrome (Congenital, familial and genetic disorders) | 1
Abdominal compartment syndrome (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Gastrointestinal oedema (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Multi-organ failure (General disorders) | 1
Pyrexia (General disorders) | 5
Hepatic failure (Hepatobiliary disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Aspergillosis (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Bronchitis viral (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urinary tract infection fungal (Infections and infestations) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Blood phosphorus decreased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Urine analysis abnormal (Investigations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Acidosis hyperchloraemic (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Unresponsive to stimuli (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Polyuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypoperfusion (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Shock (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=27)
Left atrial dilatation (Cardiac disorders) | 1
Left ventricular hypertrophy (Cardiac disorders) | 2
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 2
Vertigo (Ear and labyrinth disorders) | 1
Conjunctivitis (Eye disorders) | 1
Conjunctivitis allergic (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal pain lower (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 12
Dyspepsia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 6
Chest discomfort (General disorders) | 3
Chills (General disorders) | 2
Fatigue (General disorders) | 9
Non-cardiac chest pain (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 2
Pyrexia (General disorders) | 10
Cholelithiasis (Hepatobiliary disorders) | 1
House dust allergy (Immune system disorders) | 1
Candidiasis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 11
Oral herpes (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 2
Vulvovaginal mycotic infection (Infections and infestations) | 2
Animal bite (Injury, poisoning and procedural complications) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 2
Joint injury (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood 1,25-dihydroxycholecalciferol decreased (Investigations) | 1
Blood creatinine increased (Investigations) | 2
Ejection fraction decreased (Investigations) | 1
Electrocardiogram ST-T change (Investigations) | 2
Hepatic enzyme increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Urine albumin/creatinine ratio abnormal (Investigations) | 1
Urine albumin/creatinine ratio increased (Investigations) | 1
Urine output decreased (Investigations) | 2
Weight decreased (Investigations) | 1
Alkalosis (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Carnitine deficiency (Metabolism and nutrition disorders) | 2
Copper deficiency (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Selenium deficiency (Metabolism and nutrition disorders) | 1
Vitamin A deficiency (Metabolism and nutrition disorders) | 1
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 3
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1
Vitamin B6 deficiency (Metabolism and nutrition disorders) | 1
Vitamin C deficiency (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 5
Vitamin E deficiency (Metabolism and nutrition disorders) | 1
Zinc deficiency (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Extremity contracture (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Basal ganglion degeneration (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 9
Hypoaesthesia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Chromaturia (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Ingrown hair (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 7
Skin irritation (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3
Wisdom teeth removal (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes